CLINICAL TRIAL: NCT03353454
Title: Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat (SHP625) in the Treatment of Pediatric Subjects With Progressive Familial Intrahepatic Cholestasis (PFIC)
Brief Title: A Placebo-controlled Study of Maralixibat (SHP625) in Pediatric Subjects With Progressive Familial Intrahepatic Cholestasis (PFIC)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn due to change of ownership of the study drug maralixibat. Future studies of maralixibat will be posted by Mirum Pharmaceuticals.
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP625-306; 2017-003138-99 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-27 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Progressive Familial Intrahepatic Cholestasis (PFIC)
Keywords: Cholestasis; Maralixibat; Mutation
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Cholestasis | interventions — maralixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maralixibat (SHP625) (Experimental): Participants will be randomized to Maralixibat oral solution (up to 600 microgram per kilogram [mcg/kg]) orally twice daily for 26 weeks.
  Interventions: Drug: Maralixibat
- Placebo (Placebo Comparator): Participants will receive placebo matched to maralixibat oral solution twice daily for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maralixibat — Maralixibat oral solution (up to 600 mcg/kg) orally twice daily for 26 weeks.
  Other Names: SHP625
  Arms: Maralixibat (SHP625)
Drug: Placebo — Placebo matching to maralixibat orally twice daily for 26 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the investigational treatment (maralixibat) is safe and effective in pediatric participants with Progressive Familial Intrahepatic Cholestasis (PFIC).

ELIGIBILITY:
Key Inclusion Criteria:

* Informed consent and assent (as applicable for participants less than or equal to (<=) 18 years per Institutional Review Board/Ethics Committee (IRB)/Ethics Committee (EC) as appropriate.
* Male or female participants between the ages of 12 months and 18 years inclusive (primary cohort) or birth to 18 years inclusive (exploratory cohort) at time of consent, with a body weight greater than or equal to (>=) 5 kilogram (kg).
* Cholestasis as manifested by total sBA greater than (>) 3*upper limit of normal (ULN)
* An average AM ItchRO(Obs) score >= 1.5 during the 4 weeks leading to the baseline visit
* Diagnosis of PFIC based on:

  a. Primary cohort: i. Participants with 2 documented mutant alleles in ABCB11 (PFIC2); participants without bile salt export pump (BSEP) function (biallelic truncating mutations in ABCB11) will not be enrolled into the primary cohort. b. Exploratory cohort: i. Participants with PFIC1/3/4 or PFIC2 with biallelic truncating mutationsiii.Infants from birth to <12 months of age with PFIC ii. Participants with PFIC after internal or external (eg, PEBD) biliary diversion surgery with unsatisfactory pruritus control or where biliary diversion was reversed.

Key Exclusion Criteria:

* Chronic diarrhea requiring intravenous fluid or nutritional intervention for the diarrhea and/or its sequelae.
* History of surgical disruption of the enterohepatic circulation (applies to primary cohort only).
* Liver transplant
* Decompensated cirrhosis (international normalized ratio [INR] >1.5, albumin <30 gram per liter [g/L], history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy).
* ALT >15*ULN at screening.
* History or presence of other liver disease.
* History or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (example [eg], inflammatory bowel disease), per investigator discretion.
* Liver mass on imaging
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Any prior cancer diagnosis except for in situ carcinoma or cancers treated within 5 years of the screening visit (Visit 0) with no evidence of recurrence.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-25 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Response as Measured by the Observer Itch Reported Outcome (ItchRO[Obs]) | Baseline up to Week 26
  Compare the percentage of participants on active treatment versus (vs.) placebo who meet response criteria which is defined as improvement in before midday (AM) Observer Itch Reported Outcome (ItchRO[Obs]) severity decrease from baseline demonstrated on at least 2 of the last 3 study visits.

SECONDARY OUTCOMES:
Treatment Response as Measured by the Observer Itch Reported Outcome (ItchRO[Obs]) and Serum Bile Acids (sBA) | Baseline up to Week 26
  Compare the percentage of participants on active treatment versus (vs.) placebo who meet response criteria which is defined as improvement in average before midday (AM) Observer Itch Reported Outcome (ItchRO[Obs]) severity decrease from baseline and normalization or reduction from baseline sBA demonstrated on at least 2 of the last 3 study visits.
Normalization or Reduction From Baseline in Serum Bile Acids (sBA) | Baseline up to Week 26
  Compare the percentage of participants on active treatment vs. placebo with normalization or significant reduction from baseline in sBA.
Change Over Time in Daily Average Itch Reported Outcome (ItchRO[Obs]) Score | Baseline up to Week 26
  Change over time in daily average ItchRO scores will be reported.
Change Over Time in Before Midday (AM) Itch Reported Outcome (ItchRO[Obs]) Score | Baseline up to Week 26
  Change over time in AM ItchRO scores will be reported.
Change Over Time in After Midday (PM) Itch Reported Outcome (ItchRO[Obs]) Score | Baseline up to Week 26
  Change over time in PM ItchRO scores will be reported.
Disappearance of Pruritus as Measured by Observer Itch Reported Outcome (ItchRO[Obs]) | Baseline up to Week 26
  Compare the percentage of participants on active treatment vs. placebo of participants who experience disappearance of pruritus as measured by ItchRO(Obs).
Improvement in Height | Baseline up to Week 26
  Number of participants on active treatment vs. placebo with a height z-score change from baseline >0.
Improvement in Weight | Baseline up to Week 26
  Number of participants on active treatment vs. placebo with a weight z-score change from baseline >0.
Change From Baseline in Nutritional Status as Measured by Mid-arm Circumference | Baseline, Week 26
  Compare the change in nutritional status as measured by mid-arm circumference in participants on active treatment vs. placebo.
Change From Baseline in Nutritional Status as Measured by Triceps Skin Fold | Baseline, Week 26
  Compare the change in nutritional status as measured by triceps skin fold in participants on active treatment vs. placebo.
Change From Baseline in Clinician Scratch Scale (CSS) | Baseline, Week 26
  Compare the change in Clinician Scratch Scale score in participants on active treatment vs. placebo.
Change From Baseline in Quality of Life as Measured by Pediatric Quality of Life Inventory (PedsQL) | Baseline, Week 26
  Compare the change from baseline of PedsQL in participants on active treatment vs. placebo.
Change From Baseline in Quality of Sleep as Measured by Children's Sleep Habits Questionnaire (CSHQ) | Baseline, Week 26
  Compare the change from baseline of CSHQ in participants on active treatment vs. placebo.
Normalization or Meaningful Reduction From Baseline of Alanine Aminotransferase (ALT) | Baseline up to Week 26
  Number of participants whose ALT normalizes on treatment or has decreased >=50%.
Normalization or Meaningful Decrease From Baseline of Total Bilirubin | Baseline up to Week 26
  Number of participants whose total bilirubin normalizes on treatment or has decreased >=50%.
Change From Baseline in Biomarkers of Bile Acid Synthesis | Baseline, Week 26
  Change from baseline in biomarkers of bile acid synthesis (serum 7 alpha-hydroxy-4-cholesten-3-one [C4]).
Evaluate the safety of SHP625 | Baseline up to Week 26
  Adverse events, changes in vital signs, laboratory, and other safety parameters will be compared between participants on active treatment vs. placebo.
Plasma Levels of Maralixibat Over Time | Baseline, Week 6, 10, 14, 18, 22 and 26
  Systemic concentrations of maralixibat in plasma will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum

IPD SHARING:
Plan to Share IPD: No